CLINICAL TRIAL: NCT00006300
Title: Oral Manifestations of Aplastic Anemia
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000113; 00-D-0113
Record Dates: First submitted 2000-09-27; First posted 2000-09-28 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-04

CONDITIONS: Aplastic Anemia
Keywords: Immunosuppression; Treatment Recommendations; Pancytopenia; Schizophrenia; Inpatient Population
MeSH Terms: conditions — Anemia, Aplastic; Pancytopenia; Schizophrenia

SUMMARY:
The purposes of this study are threefold: 1) to evaluate the prevalence and risks of oral complications in patients with aplastic anemia; 2) to evaluate if oral problems in these patients can predict their response to treatment; and 3) to review complications of dental treatment in these patients in order to establish treatment guidelines.

This study will be performed through a review of medical charts of 79 patients with aplastic anemia and 67 patients with schizophrenia who were treated at the National Institutes of Health Dental Clinic between 1993 and 1999. The schizophrenia patients will serve as a control population.

Demographic, clinical and radiographic information will be collected for all patients. Additional data collected only for aplastic anemia patients will include medical therapy, disease duration, blood cell counts, oral problems that developed during treatment and treatment response.

DETAILED DESCRIPTION:
The prevalence, risk factors and significance of oral manifestations in aplastic anemia have not been well characterized. Thus, in the present study, through a retrospective chart review, we document the prevalence of oral complications in AA patients and the risks for oral manifestations in a case-control study. Schizophrenic patients represent controls. Information includes the following; demographic, clinical and radiographic information for cases and controls. Additional data collection for only AA patients includes prior medical therapy, CBC and differential, disease duration, new oral manifestations during AA treatment and medical treatment response. We determine if systemic clinical features of AA predict oral manifestations, and if oral manifestations predict treatment outcomes for AA patients. Finally complications following dental treatment are compiled and reviewed to establish initial treatment guidelines for these patients.

ELIGIBILITY:
INCLUSION CRITERIA:

Cases: All aplastic anemia patients evaluated at the NIH dental clinic for consultation between 1993-1999.

Controls: All schizophrenic patients evaluated at the NIH dental clinic for consultation between 1993-1999.

EXCLUSION CRITERIA:

Patients without the diagnosis of aplastic anemia for cases or schizophrenia for the controls.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146
Dates: Start 2000-04; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Luker J, Scully C, Oakhill A. Gingival swelling as a manifestation of aplastic anemia. Oral Surg Oral Med Oral Pathol. 1991 Jan;71(1):55-6. doi: 10.1016/0030-4220(91)90521-d. PMID 1994323
- [Background] Jones JE, Coates TD, Poland C. Dental management of idiopathic aplastic anemia: report of a case. Pediatr Dent. 1981 Sep;3(3):267-70. No abstract available. PMID 6461852
- [Background] Young NS. Acquired aplastic anemia. JAMA. 1999 Jul 21;282(3):271-8. doi: 10.1001/jama.282.3.271. No abstract available. PMID 10422997